CLINICAL TRIAL: NCT05762614
Title: Analysis of the Relationship Between Ventilatory Variability and Dyspnea in Patients Under Invasive Mechanical Ventilation During a Weaning Trial
Brief Title: Respiratory Variability and Dyspnea During Spontaneous Breathing Trial
Acronym: DYSREVA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230055
Record Dates: First submitted 2023-02-10; First posted 2023-03-09 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-02

CONDITIONS: Relationship Between Dyspnea and Ventilatory Variability
Keywords: dyspnea; Ventilatory variability; Weaning; Mechanical ventilation; Intensive care
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient on invasive mechanical ventilation able to perform a SBT
  Interventions: Other: Dyspnea assessment

INTERVENTIONS:
Other: Dyspnea assessment — Dyspnea assessment, respiratory variability, Spirometry, Electromyography

SUMMARY:
In intensive care unit, dyspnea, the distressing and fearful awareness of breathing, is frequent and harmful. To be treated, dyspnea must be detected and quantified, which is impossible in approximately 50% of patients receiving invasive mechanical ventilation. However, these non-communicative patients are exposed to the same risk factors for dyspnea as communicative patients and the impossibility to communicate a suffering increases its traumatic impact. In addition, simple therapeutic means, such as optimizing the settings of the ventilator, can significantly alleviate or even eliminate dyspnea. It is therefore particularly important to be able to detect and quantify it effectively. The Mechanical Ventilation - Respiratory Distress Observation Scale (MV-RDOS) is an observational dyspnea scale that bypasses patient involvement and represents a promising tool in the detection of dyspnea in non-communicative patients. However, its use is partly based on the observation of the facial expression of fear or the abdominal paradox, the assessment of which remains subjective. The analysis of ventilatory variability, which reflects the load-capacity balance of the respiratory system, could provide an alternative to detect dyspnea in these patients. The investigators are therefore going to measure the ventilatory variability using the thoracic motion signals obtained with a force sensor integrated in a chest strap and the ventilatory flows at airways in patients receiving invasive mechanical ventilation during a spontaneous breathing trial and compare the indices of ventilatory variability with the dyspnea visual analog scale in communicative patients and with the MV-RDOS in all patients (communicative and non-communicative).

DETAILED DESCRIPTION:
1. Types of measures and techniques used 1.1. Dyspnea The presence of dyspnea will be defined by a positive response to at least 2 of the following questions: "Do you feel out of breath? " ; "Do you feel a lack of air? " ; "Is your breathing difficult? " ; "Are you having trouble breathing? ". The intensity of dyspnea will be measured by VAS-D in communicative patients. Dyspnea VAS will be used to define patients with clinically significant dyspnea (D-VAS > 30 mm) or non-clinically significant dyspnea (D-VAS ≤ 30 mm). The measurement of dyspnea by the MV-RDOS scale will be performed in all patients and clinically significant dyspnea will be strongly suspected by the value of the MV-RDOS ≥ 2.6.

1.2. Ventilatory variability

The variability will be measured from raw airway flow (reference method) and using a force sensor integrated in a chest strap. The good correlation between the measurement of ventilation by a chest strap and the reference measurement has been demonstrated in healthy volunteers and in obese subjects on all the components of the spirogram: VT, TI, TE, TTOT, VT/TI and TI /TTOT. Two variability indices will be measured:

1. The coefficient of variation (CV) of chest expansion, after pre-processing by an artifact elimination algorithm, per period of 5 minutes and displayed continuously as a trend curve on a tablet connected to the sensor
2. Frequency analysis of the respiratory signal by Fast Fourier Transformation (FFT) over periods of 5 minutes and calculation of the H1/DC component.

1.3. Surface electromyography of inspiratory extra-diaphragmatic muscles The surface EMG of the extra diaphragmatic inspiratory muscles (Alae Nasi and Parasternals) will be collected via self-adhesive surface electrodes. Bilateral recording of the parasternal muscles will be performed by a pair of electrodes placed in the second intercostal space near the sternum. The recording of the Alae nasi muscles will be performed by positioning an electrode on each nostril. The electrical signals of inspiratory muscle activity will be identified using the Labchart Peak Analysis to extract the root mean square (RMS) of the EMG (RMS-EMG). This envelope of the inspiratory RMS-EMG signal will be used for the calculation of the maximum EMG amplitude (EMGmax) and its area under the curve (EMGAUC). To minimize the artifacts related to ECG activity, the parasternal EMG signal will be filtered before the RMS averaging process, using a low pass filter (50-400 Hz).

1.4. Airway flow and pressure A disposable pneumotachograph and a differential pressure sensor connected to a demodulator will be inserted in series at the proximal end of the breathing circuit between the Y-piece and the patient, allowing measurement of airway flow and pressure.

The signals will be digitized at a sampling frequency of 40 Hz. Ventilatory volumes and times (TI, TE, FR) will be measured from flow rate curves.

4.5. Result of the ventilatory bondage test (SBT) Failure of SBT is defined by the appearance and persistence for at least 5 minutes of one of the following criteria: SpO2 ≤ 90% or PaO2 ≤ 50mmHg with FiO2 ≥ 50%, PaCO2 > 50 mmHg, pH < 7.32, respiratory rate > 35/min, heart rate > 140/min, systolic blood pressure > 180 mmHg or < 90 mmHg.

2. Sequence of experimental steps Patients will be placed in a ventilatory weaning test with 0 cmH2O of pressure support and 0 cmH2O of end-expiratory pressure. A quantification of dyspnea will be performed for all patients using the MV-RDOS score and by Dyspnea VAS (D-VAS) for communicative patients before the start of SBT, every 5 minutes during SBT and at the end of SBT. Recordings of respiratory movements, airway flow, EMG and ECG will be made at the same time, per 5-minute period, 5 minutes before the start of the weaning test and during the 30-minute weaning test.

3. Statistical analyzes Based on a 50% probability of occurrence of clinically significant dyspnea (D-VAS > 30 mm) during the SBT and a decrease in VT CV from 0.25 to 0.18 in case of failure of SBT a total of 86 patients was calculated (alpha risk at 0.05, power 85%, common standard deviation at 0.12), 43 communicative patients and 43 non-communicative. It is therefore planned to include 100 patients in total, including 50 communicative patients and 50 non-communicative patients.

Comparison between the group "clinically significant dyspnea" vs. "not clinically significant" on their variability indices (CV and H1/DC) will be performed using the non-parametric Mann-Whitney test. The two groups "successful" vs. "failure" of the SBT will be compared on their variability indices (CV and H1/DC), according to the same methods. The correlations between variability indices and intensity of dyspnea and between variability indices and surface EMG will be tested using Spearman's correlation coefficient. The performance of the variability indices and the modified MV-RDOS to predict dyspnea or failure of SBT will be estimated by calculating the area under the curve of the ROC curves. An observed difference will be considered significant if the probability "p" of a type I error is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive mechanical ventilation > 48h,
2. Readiness-to-wean ability: ability defined by all of the following criteria: effective cough, no excessive tracheo-bronchial secretions, resolution of the disease that prompted the intubation, heart rate ≤ 140/min, pressure systolic blood pressure between 90 and 160 mmHg, no or very low dose of amines, SpO2 > 90% in 40% FiO2 (or PaO2/FiO2 > 150), positive expiratory pressure < 8 cmH2O, respiratory rate ≤ 35/min, tidal volume > 5ml/kg of theoretical body weight, respiratory rate / tidal volume ratio < 105 cycles/min/L
3. Decision by the clinician in charge of the patient to perform a SBT,
4. Patient or close consent obtained,
5. Person affiliated to a Social Security scheme or beneficiary (excluding AME).

Exclusion Criteria:

1. Minor patient,
2. Pregnant or breastfeeding woman,
3. Agitation/sedation: RASS > 2 or < 2,
4. Post-operative thoracic or abdominal surgery,
5. Chest skin lesion contraindicating the placement of a chest strap,
6. Person under legal protection (guardianship, curators), safeguarded by justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient on invasive mechanical ventilation able to perform a SBT
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Clinically significant dyspnea - D-VAS | during SBT
  Clinically important dyspnea defined by a Dyspnea visual analog scale (D-VAS) > 30 mm for communicating patients
Clinically significant dyspnea - MV-RDOS | during SBT
  Mechanical Ventilation Respiratory Distress Observation Scale(MV-RDOS) ≥ 2.6 for all patients

SECONDARY OUTCOMES:
Intensity of dyspnea | during SBT
  Dyspnea visual analog scale (D-VAS) values or Mechanical Ventilation Respiratory Distress Observation Scale(MV-RDOS) values
issue of the SBT | one day
  success or failure of the SBT
EMG signal | during SBT
  Maximum amplitude and area under the envelope curve of the EMG signal of the extra-diaphragmatic respiratory muscles indicating dyspnoea.

CONTACTS AND LOCATIONS:
Overall Officials: Maxens Decavele, MD, Principal Investigator — APHP
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.